CLINICAL TRIAL: NCT04094207
Title: The Phosphodiesterase Inhibitor Pentoxifylline as an Adjunctive in Treatment of Negative Symptoms in Chronic Schizophrenia: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Pentoxifylline as an Adjunctive in Treatment of Negative Symptoms in Chronic Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principal Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4/2021NEUR1
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Equivalent Placebo will be given
  Interventions: Drug: Placebo oral tablet
- Pentoxifylline group (Experimental): Pentoxifylline will be given orally at 800 mg a day for 8 weeks
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Placebo oral tablet — Placebo tablets PLUS Risperidone 2 mg tablet up to 6 mg/day
  Arms: Control group
Drug: Pentoxifylline — Pentoxifylline tablet PLUS Risperidone 2 mg tablet up to 6 mg/day
  Arms: Pentoxifylline group

SUMMARY:
The aim of this study to evaluate the efficacy and safety of pentoxifylline, the novel phosphodiesterase inhibitor, as an adjunctive to risperidone in alleviating the negative symptoms of schizophrenia.

DETAILED DESCRIPTION:
there is some evidence for the role of phosphodiesterase (PDE) signaling system in pathophysiology of schizophrenia making this system a potential target for therapeutic agents. PDEs are a family of enzymes that hydrolyse cyclic nucleotides and thus play a key role in regulating intracellular levels of the second messenger cyclic adenosine monophosphate (cAMP) and cyclic guanosine monophosphate. Pentoxifylline (PTX) is a methylated xanthine derivative and a PDE inhibitor that is FDA-approved for the treatment of patients with intermittent claudication on the basis of chronic occlusive arterial disease of the limbs. It is known to inhibit platelet aggregation, increase erythrocyte flexibility or deformability, and reduce blood viscosity. The rationale for its use in schizophrenia is that it competitively inhibits PDEs, resulting in increased cAMP levels, the activation of protein kinase A (PKA), the inhibition of IL and TNF-α synthesis, and reduced inflammation. Furthermore, there is growing evidence to support the inflammatory hypothesis of schizophrenia, the investigators will also explore whether cytokine levels mediate the response from pentoxifylline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-40 years
* Males & females
* patients between the ages of 18 and 53 who met the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (20), with a minimum disease duration of two years.
* stable on risperidone for a minimum of 8 weeks
* clinically stable for at least 4 weeks prior to study.
* willing to give informed consent.
* able to take medication orally.

Exclusion Criteria:

* Acute, unstable, significant or untreated medical illness beside schizophrenia;
* Pregnant or breast-feeding females;
* History of substance abuse or dependence in the past 3 months.
* Known contraindication to pentoxifylline treatment.
* Any serious or life-threatening medical conditions or neurological problem, severe extrapyramidal symptoms, history of abnormal bleeding, presence of hypothyroidism, renal disease, cardiovascular problems, rising liver transaminases to 3 times the upper limit of normal or higher

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment-induced change in total score on Positive and Negative Syndrome Scale (PANSS) | Baseline to week 8 of the study
  PANSS total score will be used to examine treatment-induced change in psychaopthology. The PANSS is a 30-item rating scale used to assess symptoms of psychopathology. We will use the total PANSS score as the primary outcome measure which reflects total level of psychopathology including the positive and negative symptoms as well as general psychopathology.This measure will be administered at baseline, week 8 and week 16 of the study to assess if pentoxifylline treatment results in a significant reduction in PANSS total score as opposed to placebo.

SECONDARY OUTCOMES:
Treatment-induced changes in plasma level of cytokines | Baseline and week 8 of the study
  Cytokine levels will assessed at baseline and week 8 of the study to examine treatment-induced changes in neuroinflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Abdallah MS, Mosalam EM, Hassan A, Ramadan AN, Omara-Reda H, Zidan AA, Samman WA, El-Berri EI. Pentoxifylline as an adjunctive in treatment of negative symptoms in chronic schizophrenia: A double-blind, randomized, placebo-controlled trial. CNS Neurosci Ther. 2023 Jan;29(1):354-364. doi: 10.1111/cns.14010. Epub 2022 Nov 7. PMID 36341700